CLINICAL TRIAL: NCT02693405
Title: Assessment of Executive and Socio-cognitive Functions in Child and Adult Survivors of Primary Brain Tumor: Impact on Patients' and Relatives' Quality of Life.
Brief Title: Executive and Socio-cognitive Functions in Survivors of Primary Brain Tumor: Impact on Patients' Quality of Life
Acronym: NEUROCOG-QOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-P2015-06
Record Dates: First submitted 2016-02-05; First posted 2016-02-26 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Primary Brain Tumor; Neurocognition; Quality of Life
MeSH Terms: conditions — Brain Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- child and adult survivors of brain tumor (Experimental): Executive functions and social cognition will be assessed using cognitive (Stroop task, Modified Card Sorting Task, Digit spans) and behavioral (BRIEF for childrens and BRIEF-A for adults) tests.
  Quality of life will be assessed by questionaires (SF-36, QLQC30-BN20 for adults and Peds-Ql for childrens)
  Interventions: Other: Executive functions; Other: social cognition; Other: quality of life
- healthy controls (Experimental): Executive functions and social cognition will be assessed using cognitive (Stroop task, Modified Card Sorting Task, Digit spans) and behavioral (BRIEF for childrens and BRIEF-A for adults) tests.
  Quality of life will be assessed by questionaires (SF-36, QLQC30-BN20 for adults and Peds-Ql for childrens)
  Interventions: Other: Executive functions; Other: social cognition; Other: quality of life

INTERVENTIONS:
Other: Executive functions — measures of executive functioning with tasks
Other: social cognition — measures of socio-cognitive functioning with tasks
Other: quality of life — measures of quality of life with questionnaires

SUMMARY:
Significant advances in primary malignant brain tumors (PBT) treatment have led to dramatically improved survival, both in children and adults. However, survival has not come without a cost and aggressive treatment methods associated with significant long-term adverse effects, often referred to as "late effects" (Panigrahy & Blüml, 2009). These effects are the medical, physical, cognitive and psychosocial sequelae associated with cancer and its treatments that generally emerge two to five years after treatment ends (e.g., Landier & Bhatia, 2008).

The most serious challenge survivors of brain tumors face may be cognitive dysfunction. One especially important cognitive domain is executive functioning, which refers to essential factors such as problem-solving, goal-directed behavior and the ability to maintain stable interpersonal relationships (Lezak et al., 2004). Despite the potential impact of executive impairments on behavioral regulation and quality of life, few studies were conducted with survivors of PBT specifically for the assessment of executive functioning. Another fundamental neuro-cognitive domain is social cognition, which refers to the ability to understand the intentions and beliefs of others (Frith & Singer, 2008). Social cognitive deficits are expected to impair autonomy and relationships, but scarce attention has been devoted to the study of social cognition in survivors of PBT and no study has attempted to compare socio-cognitive data and measures of health-related quality of life. It is noteworthy that executive function and socio-cognitive skills improve throughout childhood and adolescence, and improvements in these skills have frequently been attributed to maturation of the brain, especially the prefrontal cortex (e.g., Tamnes et al., 2010). This suggests a greater impact of the disease and its treatment on these functions in children/adolescents.

DETAILED DESCRIPTION:
First, the investigators will calculate the prevalence of cognitive and socio-cognitive deficits, by comparing the performances of patients (children/adolescents and adults) to normative data available for each tasks and to performances of healthy controls matched on socio-demographic criteria.

Second, the investigators will compare the neuropsychological scores for cognitive and socio-cognitive tasks to health related quality of life (HRQOL) data (composite scores and by domains). Comparisons of neuropsychological and HRQOL scores will be performed between the two populations (children / adolescents and adults).

Third, the investigators will compare the data from the two age groups for the aforementioned variables (cognitive and behavioral executive assessments, cognitive and affective TOM). The proximity of the tasks should provide valid elements of comparison. The investigators will compare the questionnaires in auto-and hetero-evaluation for each HRQOL scales, and also for executive behavioral questionnaires.

Finally, to evaluate the investigators will compare the HRQOL patients/relatives' data to measure the potential impact of the disease on HRQOL of relatives of PBT survivors and the potential link between these data.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 59
* Children/adolescents and adults who have been treated by chemotherapy and/or radiotherapy and/or neurosurgery, subsequent to the diagnosis of a primary brain tumor
* The end of treatment must be comprised between 2 and 5 years at the time of the assessment, as argued above.

Exclusion Criteria:

* Sensory disturbances (e.g., visual, auditory) incompatible with the achievement of the tasks
* Language or praxis deficits inconsistent with the achievement of the tasks
* Neurological disease other than PBT
* secondary brain tumor
* Psychiatric history (consultation with a psychiatrist of the University Hospital if doubt)
* Insufficient French language proficiency

Ages: 8 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
performances in executive tasks and executive questionnaires | 2 years
  Executive functions will be assessed using executive cognitive tasks (Stroop task for inhibition, Modified Card Sorting Task for mental flexibility, Digit spans for working memory) and questionnaires (BRIEF for childrens and BRIEF-A for adults) for executive behavioral measures.
  Standardized norms in French are available for these tasks, which permit determining if the performances are pathological. So, these multiple measurements will be aggregated to determine the number of patients with pathological performances for executive tasks (tasks and questionaires).
performances in social cognition tasks | 2 years
  The first task involves a mental representation or belief about the state of the world (eg, Samson, 2012). The items offered in this kind of task are used to assess the ability to understand that the belief to infer in a type of scenario does not correspond to the reality.
  The second task will be the Faux Pas task (Stone et al., 1998). This task is composed of written scenarios and the subject must detect if someone has done or said something he should not have said- the "faux pas". If the subject detects that there was a faux pas, additional questions are asked to detect whether he/she understands the cognitive side and the emotional side of the faux pas.
  Standardized norms in French are available for these tasks, which permit determining if the performances are pathological. These multiple measurements will be aggregated to determine the number of patients with pathological performances.

SECONDARY OUTCOMES:
quality of life questionnaires | 2 years
  Health-related quality of life (HRQOL) will be assessed in adults with the French validated version of the 36-Item Short Form Survey (SF-36; Ware & Sherbourne 1992) and a specific questionnaire for assessing quality of life of patients with brain tumors (QLQ-C30-BN20), commonly used in the international literature (eg, Chen et al, 2012;. Pulenzas et al, 2014).
  Regarding the HRQOL assessment in children, the choice fell on the Peds-Ql. The PEDS QL measures HRQOL with three major composite assessments -psychosocial, physical, and total HRQOL.
  Standardized norms in French are available for questionaires, which permit determining if the performances are pathological. These measurements will be aggregated to determine the number of patients with abnormal performances for these questionaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Besnard, PhD, Principal Investigator — University of Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frith CD, Singer T. The role of social cognition in decision making. Philos Trans R Soc Lond B Biol Sci. 2008 Dec 12;363(1511):3875-86. doi: 10.1098/rstb.2008.0156. PMID 18829429
- [Background] Landier W, Bhatia S. Cancer survivorship: a pediatric perspective. Oncologist. 2008 Nov;13(11):1181-92. doi: 10.1634/theoncologist.2008-0104. Epub 2008 Nov 5. PMID 18987046
- [Background] Lezak, M.D., Howieson, D.B., & Loring, D.W. (2004). Neuropsychological Assessment. New York, NY: Oxford University Press.
- [Background] Panigrahy A, Bluml S. Neuroimaging of pediatric brain tumors: from basic to advanced magnetic resonance imaging (MRI). J Child Neurol. 2009 Nov;24(11):1343-65. doi: 10.1177/0883073809342129. PMID 19841424
- [Background] Tamnes CK, Ostby Y, Walhovd KB, Westlye LT, Due-Tonnessen P, Fjell AM. Neuroanatomical correlates of executive functions in children and adolescents: a magnetic resonance imaging (MRI) study of cortical thickness. Neuropsychologia. 2010 Jul;48(9):2496-508. doi: 10.1016/j.neuropsychologia.2010.04.024. Epub 2010 Apr 29. PMID 20434470
- [Background] Caissie A, Nguyen J, Chen E, Zhang L, Sahgal A, Clemons M, Kerba M, Arnalot PF, Danjoux C, Tsao M, Barnes E, Holden L, Danielson B, Chow E. Quality of life in patients with brain metastases using the EORTC QLQ-BN20+2 and QLQ-C15-PAL. Int J Radiat Oncol Biol Phys. 2012 Jul 15;83(4):1238-45. doi: 10.1016/j.ijrobp.2011.09.025. Epub 2011 Dec 13. PMID 22172909
- [Background] Pulenzas N, Khan L, Tsao M, Zhang L, Lechner B, Thavarajah N, Barnes E, Danjoux C, Holden L, Lauzon N, Sheehan P, Bedard G, Chow E. Fatigue scores in patients with brain metastases receiving whole brain radiotherapy. Support Care Cancer. 2014 Jul;22(7):1757-63. doi: 10.1007/s00520-014-2140-4. Epub 2014 Feb 9. PMID 24510194
- [Background] Samson, D. (2012). Neuropsychologie de la théorie de l'esprit chez l'adulte : Etat de l'art et implications cliniques. In P. Allain, G. Aubin & D. L. Gall (Eds.), Cognition sociale et neuropsychologie (pp. 47-63). Marseille: Solal
- [Background] Stone VE, Baron-Cohen S, Knight RT. Frontal lobe contributions to theory of mind. J Cogn Neurosci. 1998 Sep;10(5):640-56. doi: 10.1162/089892998562942. PMID 9802997
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Derived] Cantisano N, Menei P, Roualdes V, Seizeur R, Allain P, Le Gall D, Roy A, Dinomais M, Laurent A, Besnard J. Relationships between executive functioning and health-related quality of life in adult survivors of brain tumor and matched healthy controls. J Clin Exp Neuropsychol. 2021 Dec;43(10):980-990. doi: 10.1080/13803395.2022.2040432. Epub 2022 Mar 1. PMID 35230209